CLINICAL TRIAL: NCT00199823
Title: Autologous Stem Cell Transplantation in Acute Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Ullevaal University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-03115
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2010-09

CONDITIONS: Acute Anterior Wall Myocardial Infarction
Keywords: Myocardial infarction; bone marrow cells; cell transplantation
MeSH Terms: conditions — Anterior Wall Myocardial Infarction; Myocardial Infarction

INTERVENTIONS:
Genetic: Intracoronary aotologous stem cell transplantation

SUMMARY:
Objectives

Intracoronary transplantation of different cell populations have been used in acute myocardial infarction (AMI) with promising results. The primary objective of the ASTAMI study is to test whether intracoronary transplantation of autologous mononuclear bone marrow cells (mBMC) improve left ventricular ejection fraction (LVEF) after anterior wall AMI.

Design

The ASTAMI study is a randomized, controlled, prospective study. One hundred patients with acute anterior wall ST-elevation myocardial infarction (STEMI) treated with acute PCI are randomized in a 1:1 way to either intracoronary transplantation of autologous mBMC 5-8 days after PCI or to control. Left ventricular function, exercise capacity, biochemical status, functional class, quality of life and complications are validated at baseline and during a 12-month follow up.

ELIGIBILITY:
Inclusion criteria:

* age 40-75 years
* anterior wall AMI with 120-720 minutes from onset of symptoms to PCI
* ST elevation on ECG according to WHO criteria
* angiographically significant stenosis on LAD proximal to the second diagonal branch
* successful PCI with stenting of culprit lesion
* hypokinetic, akinetic or dyskinetic segments assessed by echocardiography in a standard 16 segment model and
* CK-MB above 3 times upper reference value.

Exclusion criteria:

* previous MI with established significant Q-waves on ECG
* cardiogenic shock
* permanent pacemaker or other contraindication to MRI
* stroke with significant sequela
* short life expectancy due to extra cardiac reason
* uncontrolled endocrinological disturbance
* HIV and/or HBV/HCV positive serology
* mental disorder or other condition which interferes with patient possibility to comply with the protocol.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-09; Study Completion 2006-05

PRIMARY OUTCOMES:
whether intracoronary mBMC transplantation improve LVEF after AMI assessed by ECG-gated SPECT.

SECONDARY OUTCOMES:
To test whether mBMC treatment improve exercise capacity assessed by bicycle ergometry
To test whether mBMC treatment improve quality of life assessed by the SF 36 formula

CONTACTS AND LOCATIONS:
Overall Officials: Ketil Lunde, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Norway

REFERENCES:
- [Result] Lunde K, Solheim S, Aakhus S, Arnesen H, Abdelnoor M, Egeland T, Endresen K, Ilebekk A, Mangschau A, Fjeld JG, Smith HJ, Taraldsrud E, Grogaard HK, Bjornerheim R, Brekke M, Muller C, Hopp E, Ragnarsson A, Brinchmann JE, Forfang K. Intracoronary injection of mononuclear bone marrow cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1199-209. doi: 10.1056/NEJMoa055706. PMID 16990383
- [Derived] Solheim S, Seljeflot I, Lunde K, Bratseth V, Aakhus S, Forfang K, Arnesen H. The influence of intracoronary injection of bone marrow cells on prothrombotic markers in patients with acute myocardial infarction. Thromb Res. 2012 Nov;130(5):765-8. doi: 10.1016/j.thromres.2011.11.045. Epub 2011 Dec 20. PMID 22192151
- [Derived] Hopp E, Lunde K, Solheim S, Aakhus S, Arnesen H, Forfang K, Edvardsen T, Smith HJ. Regional myocardial function after intracoronary bone marrow cell injection in reperfused anterior wall infarction - a cardiovascular magnetic resonance tagging study. J Cardiovasc Magn Reson. 2011 Mar 17;13(1):22. doi: 10.1186/1532-429X-13-22. PMID 21414223